CLINICAL TRIAL: NCT03617068
Title: The Effectiveness and Dermato-pharmacokinetic of Coconut Oil Cream as a Prevention Treatment for Occupational Hand Dermatitis Among Batik Workers
Brief Title: The Effectiveness of Coconut Oil Cream as a Prevention Treatment for Occupational Hand Dermatitis Among Batik Workers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 05
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-06

CONDITIONS: Hand Dermatoses
MeSH Terms: conditions — Hand Dermatoses

STUDY DESIGN:
Intervention Model Description: Batik traditional workers with occupational hand dermatitis using emolient for prevention
Who Masked: Participant, Investigator
Masking Description: blinding had to be done by Clinical Research Supporting Unit Faculty of Medicine, Universitas Indonesia
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coconut Oil Cream (Active Comparator): This group consist of batik traditional workers who use coconut oil cream for 2 weeks.
  Interventions: Drug: Cocos Nucifera Whole
- Placebo Cream (Placebo Comparator): This group consist of batik traditional workers who use placebo cream which contained the vehiculum of the cream; using for 2 weeks.
  Interventions: Drug: Cocos Nucifera Whole

INTERVENTIONS:
Drug: Cocos Nucifera Whole — Applying the Cocos Nucifera Whole cream for 2 weeks, on both of arms. We evaluated the score of hand dermatitis using Hand Eczema Score Index ( HECSI), transepidermal water loss (TEWL), and Skin capacitance
  Other Names: Coconut Oil Cream
Drug: Cocos Nucifera Whole — For dermatopharmacokinetic evaluation using tape/ skin stripping
  Other Names: Coconut Oil Cream

SUMMARY:
Empirically, mosturizer is used to prevent and treat many occupational dermatoses that has skin barrier impairment. Evidence based medicine about the effectivity of mosturizer in occupational dermatoses is limited. Coconut oil is one of traditional substance that is used as a skin care. There is study shows that coconut oil is effective for atopic dermatitis treatment in children. Other studies are needed to assess the effectivity coconut oil mosturizer cream to overcome occupational hand dermatitis.

DETAILED DESCRIPTION:
The aim of this study is to measure the effectivenes of coconut oil cream for batik workers who suffer from occupational hand dermatitis. The gloves that used as a protective equipment are made from rubber which have its own limitations. Therefore other interventions are needed to improve barrier skin.

ELIGIBILITY:
Inclusion Criteria:

* signing the informed consent document before the study start
* adult population include patients between the ages of 18 and 64 years who work in the dyeing and washing process more than 6 months.
* suffering from occupational hand dermatitis that meet Mathias Criteria.
* willing to obey the research protocol
* willing to fill in diary periodically

Exclusion Criteria:

* having history of allergy or irritation caused by coconut oil or other mosturizer
* suffering from symptoms including edema, exudation, crust, fissures, liver problems, and signs of infection
* on corticosteroid treatment ( medium to high potency) or on systemic immunosuppressive therapy

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
clinical improvement of hand dermatitis measured by Hand Eczema Severity Index (HECSI) after using coconut oil | 14 days
  Batik workers who had hand dermatitis was measured using HECSI score before and after intervention with coconut oil cream. They used the cream twice daily for 14 days

SECONDARY OUTCOMES:
Transepidermal water loss (TEWL) | 14 days
  TEWL is the amount of water that passively evaporates through skin to the external environment
Skin capacitance | 14 days
  Skin capacitance depends on the water content of the stratum corneum

CONTACTS AND LOCATIONS:
Overall Officials: Retno W Soebaryo, Prof, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data